CLINICAL TRIAL: NCT04973540
Title: A Prospective, Multi-center, Single-arm Clinical Trial to Evaluate the Safety and Efficacy of Iron Bioresorbable Scaffold System (IBS Angel) in Patients With Pulmonary Artery Stenosis
Brief Title: A Clinical Trial to Evaluate the Safety and Efficacy of IBS Angel in Patients With Pulmonary Artery Stenosis
Acronym: IRIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biotyx Medical (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBS Angel-01
Record Dates: First submitted 2021-06-11; First posted 2021-07-22 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Pulmonary Artery Stenosis
MeSH Terms: conditions — Stenosis, Pulmonary Artery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBS Angel (Experimental): Iron Bioresorbable Scaffold System
  Interventions: Device: Iron Bioresorbable Scaffold System (IBS Angel)

INTERVENTIONS:
Device: Iron Bioresorbable Scaffold System (IBS Angel) — Subjects in this arm will be implanted with IBS Angel.

SUMMARY:
This is a prospective, multi-center, single-arm clinical trial to evaluate the safety and efficacy of Iron Bioresorbable Scaffold System (IBS Angel) in patients with pulmonary artery stenosis.

DETAILED DESCRIPTION:
82 patients with pulmonary artery stenosis will be treated with the Iron Bioresorbable Scaffold System (IBS Angel) developed by Biotyx Medical (Shenzhen) Co., Ltd. This study is designed as a prospective, multi-center, single-arm clinical trial. Enrolled patients will undergo IBS Angel implantation and will be followed up at 1, 3, 6, 12, and 24 months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must between 1 and 14 years old.
2. Patients who have congenital or secondary pulmonary artery stenosis (including pulmonary artery trunk, left pulmonary artery and right pulmonary artery), and meeting one of the following criteria:

   A: The pressure gradient across the stenosis ≥20mmHg measured by catheter; B: The degree of pulmonary artery stenosis ≥50% ( calculated by (diameter of adjacent normal segments - residual lumen diameter of the stenosis segment)/diameter of adjacent normal segments ×100%); C: The ratio of right ventricular systolic pressure to aortic systolic pressure ≥50%.
3. Patients and whose family have high compliance, voluntarily participate in and sign the informed consent form, and complete the 2-year follow-up.
4. Patients have life expectancy >2 year after successful stent implantation.

Exclusion Criteria:

1. Patients who have a history of disease related to iron overload or iron disorder, such as hereditary hemochromatosis, etc.
2. Patients with cardiopulmonary function that cannot tolerate surgery, such as severe heart failure (NYHA Grade III and above) that cannot be controlled by active medical treatment.
3. Patients with known allergy to contrast agent, iron and its degradation products.
4. Patients with hemorrhagic disorders.
5. Patients with contraindications on antiplatelet agents and anticoagulant therapy.
6. Patients with thrombosis at the vascular wall of target lesion or the distal or proximal location.
7. Patients with known severe renal or hepatic insufficiency which are unsuitable for index procedure as per investigator judgement.
8. Previous stent implantation has been performed to treat the target lesion;
9. Patients with severe stenosis or excessive tortuosity in the targeted vessels, or anatomical abnormalities, making it difficult for device to reach the target lesion.
10. Other conditions that are not suitable for stent delivery or balloon expansion.
11. Patient who have already participated in another drug or medical device clinical trial that have not yet completed or withdrawn within 3 months before the screening period of this trial.
12. Patients who are not suitable for participating the trial as per investigator judgement.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Estimated)
Dates: Start 2021-07-13 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rate of freedom from in-stent restenosis | 12 months
  Defined on a per target lesion basis.
Rate of procedural success | Immediately post-procedure
  Defined on a per target lesion basis.

SECONDARY OUTCOMES:
Rate of technical success | Immediately post-procedure
  Defined on a per target lesion basis.
Rate of freedom from in-stent restenosis | 1 month
  Defined on a per target lesion basis.
Rate of freedom from in-stent restenosis | 3 months
  Defined on a per target lesion basis.
Rate of freedom from in-stent restenosis | 6 months
  Defined on a per target lesion basis.
Rate of device-related adverse events | 1 month
Rate of device-related serious adverse events | 1 month
Rate of device-related adverse events | 3 months
Rate of device-related serious adverse events | 3 months
Rate of device-related adverse events | 6 months
Rate of device-related serious adverse events | 6 months
Rate of device-related adverse events | 12 months
Rate of device-related serious adverse events | 12 months
Rate of device-related adverse events | 24 months
Rate of device-related serious adverse events | 24 months
Rate of unplanned surgery or re-intervention | 1 month
Rate of unplanned surgery or re-intervention | 3 months
Rate of unplanned surgery or re-intervention | 6 months
Rate of unplanned surgery or re-intervention | 12 months
Rate of unplanned surgery or re-intervention | 24 months
Rate of stent thrombosis | 1 month
Rate of stent thrombosis | 3 months
Rate of stent thrombosis | 6 months
Rate of stent thrombosis | 12 months
Rate of stent thrombosis | 24 months
Rate of all-cause death | 1 month
Rate of all-cause death | 3 months
Rate of all-cause death | 6 months
Rate of all-cause death | 12 months
Rate of all-cause death | 24 months
Rate of stent displacement | 1 month
Rate of stent displacement | 3 months
Rate of stent displacement | 6 months
Rate of stent displacement | 12 months
Rate of adverse events | 1 month
Rate of serious adverse events | 1 month
Rate of adverse events | 3 months
Rate of serious adverse events | 3 months
Rate of adverse events | 6 months
Rate of serious adverse events | 6 months
Rate of adverse events | 12 months
Rate of serious adverse events | 12 months
Rate of adverse events | 24 months
Rate of serious adverse events | 24 months
Rate of device deficiency | Day 0

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - The Second Xiangya Hospital of Central South University, Changsha
  - Children's Hospital of Chongqing Medical University, Chongqing
  - The People's Hospital of Gaozhou, Gaozhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Fuwai Yunnan Cardiovascular Hospital, Kunming
  - Shanghai Children's Medical Center Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - General Hospital of Northern Theater Command of Chinese People's Liberation Army, Shenyang
  - Shenzhen Children's Hospital, Shenzhen
  - Fuwai Central China Cardiovascular Hospital, Zhengzhou

REFERENCES:
- [Derived] Sun L, Li JJ, Xu YK, Xie YM, Wang SS, Zhang ZW. Initial status and 3-month results relating to the use of biodegradable nitride iron stents in children and the evaluation of right ventricular function. Front Cardiovasc Med. 2022 Aug 1;9:914370. doi: 10.3389/fcvm.2022.914370. eCollection 2022. PMID 35979021